CLINICAL TRIAL: NCT06603012
Title: Behavioral Intervention for Lifestyle Physical Activity in Parkinson's Disease
Acronym: LifePD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Robert W Motl, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY2024-1038; P30AG022849 (NIH)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease (PD)
Keywords: Parkinson disease; Parkinsonian disorders; Movement disorders; Basal ganglia diseases; Brain diseases; Nervous system diseases; Central nervous system diseases; Neurodegenerative diseases; Cognition; Walking; Exercise; Physical Activity
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Movement Disorders; Basal Ganglia Diseases; Brain Diseases; Nervous System Diseases; Central Nervous System Diseases; Neurodegenerative Diseases; Motor Activity | interventions — Pliability

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GET Up PD (Experimental): Remotely-coached/guided, home-based program delivered using telerehabilitation focusing on aerobic fitness and muscle strength as a mode of training
  Interventions: Behavioral: GET Up PD
- Stretching and Flexibility (Active Comparator): Remotely-coached/guided, home-based program delivered using telerehabilitation focusing on stretching and range of motion as the mode of training
  Interventions: Behavioral: Stretching and Flexibility

INTERVENTIONS:
Behavioral: GET Up PD — * The exercise training prescription involves performing 3 days per week and include (a) aerobic exercise: 30+ minutes of moderate-intensity walking (≥100 steps/min) monitored by a waist-worn pedometer, and (b) resistance training: 1-3 sets, 8-12 repetitions of 5-10 exercises targeting lower and upper body, and core muscle groups using elastic bands.
  * Other components of the GET Up PD program include appropriate exercise equipment (pedometer, resistance bands), one-on-one coaching sessions via Zoom, action-planning via calendars, logbooks for self-monitoring, and SCT-based newsletters.
  Arms: GET Up PD
Behavioral: Stretching and Flexibility — * The training will involve the same frequency, duration, timeline, behavior change content, and interactions with behavioral coach as the GET Up PD program, and account for activity, social-contact, and attention.
  * Other components of the Stretching and Flexibility program include appropriate exercise equipment (yoga mat), one-on-one coaching sessions via Zoom, calendars, logbooks and newsletters similar to the GET Up PD program.
  Arms: Stretching and Flexibility

SUMMARY:
The investigators propose a Stage-I randomized controlled trial (RCT) of a remotely-delivered, 16-week social-cognitive theory-based behavioral intervention focusing on combined exercise (aerobic and resistance) training for yielding increases in device-measured physical activity and improvements in cognitive function, symptoms, and quality of life (QOL), and social-cognitive theory (SCT) outcomes among physically inactive persons with Parkinson's disease (PD). Participants (N=50) will be randomly assigned into exercise training (combined aerobic and resistance exercise) condition or active control (flexibility and stretching) condition. The 16-week intervention will be delivered and monitored remotely within a participant's home/community and supported by Zoom-based chats guided by SCT via a behavioral coach. Participants will receive training materials (e.g., prescriptive manual and exercise equipment), one-on-one coaching, action-planning via calendars, self-monitoring via logs, and SCT-based newsletters. The investigators hypothesize that the home-based exercise intervention will yield improvements in cognitive, symptomatic, and QOL outcomes.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder of the dopamine-producing nerve cells in the basal ganglia, and age is a primary risk factor for PD. Cognitive impairment is prevalent, disabling, and poorly managed among the 1 million adults living with PD in the United States. Indeed, cognitive impairment begins early in PD, and dementia develops in 80% of persons with PD. Cognitive impairment is further associated with worse fatigue, depression, anxiety, pain, and quality of life (QOL) in PD. Those observations underscore the importance of identifying efficacious approaches for managing cognitive impairment and its consequences, and promoting additional health benefits among those with PD. To date, researchers have examined the benefits of supervised, structured exercise training for managing outcomes of PD, but this approach has clear barriers associated with travel, transportation, and participation (i.e., loss of driving ability, social isolation, and lack of community integration) that are common in PD. The investigators believe that there is merit in the promotion of physical activity for managing cognitive dysfunction and other symptom and QOL outcomes in PD. The investigators offer a novel and innovative approach for promotion of physical activity in PD based on their extensive experiences from Phase I, II, and III randomized controlled trials (RCTs). Those RCTs indicate that the remotely-delivered, social-cognitive theory-based behavioral intervention has successfully increased self-reported and device-measured physical activity in persons with multiple sclerosis (MS). This approach has further resulted in improvements in cognition and walking outcomes, symptoms of fatigue, depression, anxiety, and pain, and QOL among persons with MS. The investigators leverage their experiences and preliminary results in MS, and propose a Stage-I RCT that examines the feasibility and efficacy of a remotely-delivered, theory-based behavioral intervention focusing on combined exercise (aerobic and resistance) training for yielding immediate improvements in device-measured physical activity (primary outcome) among persons with PD who are physically inactive. The investigators further examine the efficacy of this behavioral intervention for improvements in cognitive function, symptoms, and QOL (secondary outcomes). The proposed study, if successful, will provide experiences and pilot data necessary for the design of a subsequent Stage-II RCT that examines the efficacy of the behavioral intervention for immediate and sustained improvements of outcomes in an appropriately-powered and clearly-demarcated sample of adults with PD (i.e., those 50+ years of age who are prescreened for cognitive impairment). This line of research may yield "real-world" guidelines for physical activity that can be implemented for the treatment of cognitive dysfunction and other outcomes in PD. Such an opportunity for rehabilitation of cognitive function using an approach with broad reach and scalability is paramount considering the prevalent, disabling, and poorly managed nature of cognitive impairment in PD and limited efficacious resources for its treatment.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of PD
* Internet and email access
* willingness to complete the cognitive assessments and questionnaires, wear the accelerometer, and undergo randomization
* insufficient physical activity (i.e., not meeting current physical activity guidelines) based on a health contribution score of less than 14 units from the Godin Leisure-Time Exercise Questionnaire
* self-reported ability to ambulate without assistance
* age of 50+ years
* English as a primary language
* asymptomatic (i.e., one or fewer affirmatives on the Physical Activity Readiness Questionnaire [PAR-Q]) or physician approval for undertaking exercise training for those with 2 or more affirmatives on the PAR-Q

Exclusion Criteria:

* above inclusion criteria not met
* moderate or high risk of contraindications for possible injury or death when undertaking strenuous or maximal exercise using the PAR-Q
* severe cognitive impairment that might preclude compliance with the conditions based on a modified Telephone Interview for Cognitive Status (TICS-M) score of less than 18
* normal cognitive impairment based on the Montreal Cognitive Assessment (MoCA) score of 26 or more for avoiding ceiling effects involving change in cognitive function

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | Changes in time spent in light physical activity from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  ActiGraph Gt3X+ accelerometer; minutes spent in light physical activity per day
Physical Activity | Changes in time spent in moderate-to-vigorous physical activity from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  ActiGraph Gt3X+ accelerometer; minutes spent in moderate-to-vigorous physical activity per day

SECONDARY OUTCOMES:
Cognitive Function | Changes in SCOPA-Cog Baseline (pre-intervention) to after 16 weeks (post-intervention)
  SCales for Outcomes in PArkinson's disease - COGnition (SCOPA-Cog); scores range between 0-43, higher scores indicate better cognitive function
Fatigue Severity | Changes in fatigue severity scores from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Fatigue Severity Scale (FSS); scores range between 1 (min) and 7 (max), higher scores reflect greater fatigue severity
Depressive Symptoms | Changes in depressive symptoms scores from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms
Fatigue Impact | Changes in fatigue impact scores from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Modified Fatigue Impact Scale (MFIS); scores range between 0 (min) and 84 (max), higher scores reflect a greater impact of fatigue on daily life
Anxiety | Changes in anxiety scores from Baseline (pre-intervention) to after 16 weeks (post-intervention
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms
Perceived Pain | Changes in perceived pain from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Short-form McGill Pain Questionnaire (SF-MPQ); scores range between 0 and 45, higher scores indicate more perceived pain
Health-related Quality of Life | Changes in SF-36 scores from Baseline (pre-intervention), after 16 weeks (post-intervention)
  Short Form Health Status Survey (SF-36); scores range between 0 (min) and 100 (max), higher scores indicate better physical and mental aspects of quality of life

OTHER OUTCOMES:
Social Cognitive Theory | Changes in exercise self-efficacy from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Exercise Self-Efficacy Scale (EXSE); scores range between 0 (not at all confident) to 100 (completely confident), higher scores indicate more self-efficacy
Social Cognitive Theory | Changes in barriers for self-efficacy from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Barriers for Self-Efficacy Scale (BARSE); scores range between 0 (Not at all confident) to 100 (Completely confident), higher scores indicate more self-efficacy to overcome barriers to exercise
Social Cognitive Theory | Changes in exercise goal setting from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Exercise Goal Setting (EGS); scores range between 0 and 50, higher scores indicate stronger tendency to set goals
Social Cognitive Theory | Changes in exercise planning from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Exercise Planning (EPS); scores range between 0 and 50, higher scores indicate stronger tendency to make plans to engage in exercise and physical activity
Social Cognitive Theory | Changes in outcome expectations from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Multidimensional Outcome Expectations for Exercise Scale (MOEES), higher scores indicate greater perceptions of positive benefits of regular exercise and physical activity
Social Cognitive Theory | Changes in perceived social support for self-efficacy from Baseline (pre-intervention) to after 16 weeks (post-intervention)
  Social Provisions Scale (SPS); scores range between 6 and 24, higher scores indicate more perceived support

CONTACTS AND LOCATIONS:
Overall Officials: Robert Motl, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No